CLINICAL TRIAL: NCT04035564
Title: Early Sodium Intake in Preterm Newborns; Randomized Clinical Trial
Brief Title: Early Sodium Intake in Preterm Newborns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital del Niño "Dr. Federico Gomez Santos" (Other)
Responsible Party: Principal Investigator, csanchezg, Pediatric Nephrology, Hospital del Niño "Dr. Federico Gomez Santos"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01/03/18N01
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Hyponatremia; Premature
Keywords: Preterm infant; Sodium; Hyponatremia
MeSH Terms: conditions — Hyponatremia; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium < 1mEq/kg/day (Active Comparator): Sodium administration enteral and/or parenteral less than 1mEq/kg/day started on day of life one
  Interventions: Drug: Sodium < 1mEq/kg/day
- Sodium 5mEq/kg/day (Experimental): Sodium administration enteral and/or parenteral 5mEq/kg/day started on day of life one
  Interventions: Drug: Sodium 5mEq/kg/day

INTERVENTIONS:
Drug: Sodium < 1mEq/kg/day — Sodium administration enteral and/or parenteral less than 1mEq/kg/day started on day of life 1
  Arms: Sodium < 1mEq/kg/day
Drug: Sodium 5mEq/kg/day — Sodium administration enteral and/or parenteral 5mEq/kg/day started on day of life 1
  Arms: Sodium 5mEq/kg/day

SUMMARY:
Hyponatremia is a common complication among preterm infants, renal losses of sodium contribute to the development of hyponatremia in preterm newborns. Sodium imbalances impact in newborns outcome. There is controversy about the time of initiation and the requirements of sodium in premature infants. Hypothesis: early (24 hours of life) sodium supplementation (5mEq/kg/day) prevents the develop of hyponatremia in preterm infants.

DETAILED DESCRIPTION:
This study is a randomized controlled trial in infants less than 35 weeks gestation admitted to the Newborn Intensive Care Unit at Children Hospital in Saltillo Coahuila Mexico.

Infants receive at 24 hours of life; sodium (5mEq/kg/day) versus less than 1mEq/kg/day. Weight, serum and urine sodium, serum chloride, serum and urine creatinine, serum chloride, bicarbonate and glucose are monitored daily during the first 3 days of life. Patients are assessed for hyponatremia, hypernatremia, weight change, sepsis, necrotizing enterocolitis and intraventricular hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <35 Weeks gestation

Exclusion Criteria:

* Urinary malformations
* Congenital abdominal wall defect
* Intestinal atresia / obstruction
* Congenital heart defect

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanchez, MD, Principal Investigator — Pediatric Nephrology; Ben D Valdes, MD, Principal Investigator — Neonatology
Locations (1):
- Hospital del Niño Dr Federico Gomez Santos, Saltillo, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang J, Xu E, Xiao Y. Isotonic versus hypotonic maintenance IV fluids in hospitalized children: a meta-analysis. Pediatrics. 2014 Jan;133(1):105-13. doi: 10.1542/peds.2013-2041. Epub 2013 Dec 30. PMID 24379232
- [Background] Bhatia J. Fluid and electrolyte management in the very low birth weight neonate. J Perinatol. 2006 May;26 Suppl 1:S19-21. doi: 10.1038/sj.jp.7211466. PMID 16625217
- [Background] Moritz ML, Ayus JC. Hyponatremia in preterm neonates: not a benign condition. Pediatrics. 2009 Nov;124(5):e1014-6. doi: 10.1542/peds.2009-1869. Epub 2009 Oct 26. No abstract available. PMID 19858147
- [Background] Balasubramanian K, Kumar P, Saini SS, Attri SV, Dutta S. Isotonic versus hypotonic fluid supplementation in term neonates with severe hyperbilirubinemia - a double-blind, randomized, controlled trial. Acta Paediatr. 2012 Mar;101(3):236-41. doi: 10.1111/j.1651-2227.2011.02508.x. Epub 2011 Nov 19. PMID 22040311
- [Background] Al-Dahhan J, Haycock GB, Nichol B, Chantler C, Stimmler L. Sodium homeostasis in term and preterm neonates. III. Effect of salt supplementation. Arch Dis Child. 1984 Oct;59(10):945-50. doi: 10.1136/adc.59.10.945. PMID 6497431
- [Background] Gawlowski Z, Aladangady N, Coen PG. Hypernatraemia in preterm infants born at less than 27 weeks gestation. J Paediatr Child Health. 2006 Dec;42(12):771-4. doi: 10.1111/j.1440-1754.2006.00975.x. PMID 17096711
- [Background] Lonnqvist PA. III. Fluid management in association with neonatal surgery: even tiny guys need their salt. Br J Anaesth. 2014 Mar;112(3):404-6. doi: 10.1093/bja/aet436. Epub 2013 Dec 23. No abstract available. PMID 24368557
- [Background] Oh W. Fluid and electrolyte management of very low birth weight infants. Pediatr Neonatol. 2012 Dec;53(6):329-33. doi: 10.1016/j.pedneo.2012.08.010. Epub 2012 Oct 12. PMID 23276435
- [Background] Hartnoll G, Betremieux P, Modi N. Randomised controlled trial of postnatal sodium supplementation on oxygen dependency and body weight in 25-30 week gestational age infants. Arch Dis Child Fetal Neonatal Ed. 2000 Jan;82(1):F19-23. doi: 10.1136/fn.82.1.f19. PMID 10634836
- [Background] Hartnoll G, Betremieux P, Modi N. Randomised controlled trial of postnatal sodium supplementation on body composition in 25 to 30 week gestational age infants. Arch Dis Child Fetal Neonatal Ed. 2000 Jan;82(1):F24-8. doi: 10.1136/fn.82.1.f24. PMID 10634837
- [Background] Lorenz JM, Kleinman LI, Kotagal UR, Reller MD. Water balance in very low-birth-weight infants: relationship to water and sodium intake and effect on outcome. J Pediatr. 1982 Sep;101(3):423-32. doi: 10.1016/s0022-3476(82)80078-4. PMID 7050331
- [Background] Costarino AT Jr, Gruskay JA, Corcoran L, Polin RA, Baumgart S. Sodium restriction versus daily maintenance replacement in very low birth weight premature neonates: a randomized, blind therapeutic trial. J Pediatr. 1992 Jan;120(1):99-106. doi: 10.1016/s0022-3476(05)80611-0. PMID 1731034
- [Background] Koletzko B, Goulet O, Hunt J, Krohn K, Shamir R; Parenteral Nutrition Guidelines Working Group; European Society for Clinical Nutrition and Metabolism; European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN); European Society of Paediatric Research (ESPR). 1. Guidelines on Paediatric Parenteral Nutrition of the European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) and the European Society for Clinical Nutrition and Metabolism (ESPEN), Supported by the European Society of Paediatric Research (ESPR). J Pediatr Gastroenterol Nutr. 2005 Nov;41 Suppl 2:S1-87. doi: 10.1097/01.mpg.0000181841.07090.f4. No abstract available. PMID 16254497
- [Background] Bolisetty S, Osborn D, Sinn J, Lui K; Australasian Neonatal Parenteral Nutrition Consensus Group. Standardised neonatal parenteral nutrition formulations - an Australasian group consensus 2012. BMC Pediatr. 2014 Feb 18;14:48. doi: 10.1186/1471-2431-14-48. PMID 24548745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 30, 2018 - February 28, 2020
  Inclusion Criteria:
  * Preterm infants <35 Weeks gestation, less than 24 hrs of age.
  Exclusion Criteria:
  * Urinary malformations
  * Congenital abdominal wall defect
  * Intestinal atresia / obstruction
  * Congenital heart defect
  Location: Neonatology (Pediatric Hospital)
Period: Overall Study
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Started | 27 | 25
Completed | 23 | 19
Not Completed | 4 | 6
Not completed — Protocol Violation | 1 | 2
Not completed — No laboratory available | 2 | 2
Not completed — Guardian declined consent | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational Age (Weeks)
  Weeks | 32 (2.067) | 32.05 (2.460) | 32.02 (2.225)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 19 | 42
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 23 | 19 | 42
Birth weight [Mean (Standard Deviation); unit: Grams] | 1551.08 (447.73) | 1609.47 (394.92) | 1577.50 (420.59)
Length of hospital stay [Mean (Standard Deviation); unit: Days] — Population: Only patients who were discharged to home were included.
  Days
    number analyzed (Participants) | 16 | 14 | 30
    (all) | 28.43 (16.28) | 24.07 (18.39) | 26.40 (17.13)

OUTCOME MEASURES:

1. Primary Outcome: Hyponatremia
Description: serum sodium <130mEq/L
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Participants | 6 | 1
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.71, Chi-squared; Risk Ratio (RR) = 0.20, 95% CI 2-sided [0.026 to 1.533]

2. Primary Outcome: Hypernatremia
Description: serum sodium >150mEq/L
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Participants | 1 | 1
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.89, Chi-squared; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.081 to 18.09]

3. Secondary Outcome: % Weight Change
Description: The difference between initial weight and 72hrs weight, expressed in percentage of birth weight.
Time Frame: Initial weight (baseline) vs 72 hours
Measure: Mean (Standard Deviation); unit: % of birth weight
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
% of birth weight | -9.206 (4.305) | -6.345 (3.951)
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.032, t-test, 2 sided; Mean Difference (Final Values) = -2.861, 95% CI 2-sided [-5.461 to -0.261], Standard Error of Mean 1.286
Statistical Analysis 2: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.032, ANOVA; Mean Difference (Final Values) = -2.86, 95% CI 2-sided [-5.461 to -0.261], Standard Error of Mean 1.286

4. Secondary Outcome: Change in Serum Sodium
Description: The difference between current serum sodium and initial serum sodium
Time Frame: Initial serum sodium (baseline) vs 72 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
mEq/L | 1.921 (7.70) | 5.71 (7.05)
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.107, t-test, 2 sided; Mean Difference (Final Values) = -3.788, 95% CI 2-sided [-8.43 to 0.858], Standard Error of Mean 2.299
Statistical Analysis 2: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.107, ANOVA; Mean Difference (Final Values) = -3.78, 95% CI 2-sided [-8.43 to 0.85], Standard Error of Mean 2.299

5. Secondary Outcome: Weight Change
Description: The difference between current weight and initial weight
Time Frame: Initial weight (baseline) vs 72 hours
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Grams | -135.43 (57.46) | -96.05 (53.11)
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.028, t-test, 2 sided; Mean Difference (Final Values) = -39.38, 95% CI 2-sided [-74.18 to -4.57], Standard Error of Mean 17.22
Statistical Analysis 2: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.028, ANOVA; Mean Difference (Final Values) = -39.38, 95% CI 2-sided [-74.18 to -4.57], Standard Error of Mean 17.22

6. Secondary Outcome: Number of Participants With Late-onset Sepsis
Description: Positive blood culture and/or 5 days of continuous antimicrobial therapy
Time Frame: Patients will be followed during hospitalization, an expected average of 3 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Participants | 8 | 5
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.55, Chi-squared; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.296 to 1.932]

7. Secondary Outcome: Number of Participants With Necrotizing Enterocolitis
Description: Number of patients with Bell stage II or greater necrotizing enterocolitis
  Bell's Staging:
  Stage II A:
  Gastrointestinal signs: Increasing gastric aspirates, mild abdominal distention, fecal occult blood, absent bowel sounds.
  Systemic signs: Temperature instability, apnea, bradycardia, lethargy. Radiological findings: Intestinal dilatation, ileus, pneumatosis intestinalis.
  Stage II B:
  Gastrointestinal signs: As stage IIA plus abdominal tenderness. Systemic signs: As stage IIA plus metabolic acidosis and thrombocytopenia. Radiological findings: As stage IIA plus portal vein gas and ascites.
  Stage III A:
  Gastrointestinal signs: As stage IIB plus marked abdominal tenderness and generalised peritonitis.
  Systemic signs: As stage IIB plus hypotension and severe apnea. Radiological findings: As stage IIB
  Stage III B:
  Gastrointestinal signs: As stage IIIA As stage IIIA As stage IIIA plus pneumoperitoneum
Time Frame: Patients will be followed during hospitalization, an expected average of 3 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Participants | 2 | 2
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.84, Chi-squared; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.169 to 7.096]

8. Secondary Outcome: Number of Participants With Intraventricular Hemorrhage
Description: Bleeding into the brain´s ventricular system (intracranial ultrasound).
Time Frame: Patients will be followed during hospitalization, an expected average of 3 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Participants | 6 | 4
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.70, Chi-squared; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.266 to 2.448]

9. Secondary Outcome: Mortality
Description: Death during hospitalization.
Time Frame: Patients will be followed during hospitalization, an expected average of 3 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
Number analyzed (Participants) | 23 | 19
Participants | 5 | 2
Statistical Analysis 1: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.33, Chi-squared
Statistical Analysis 2: Comparison: Sodium < 1mEq/kg/Day vs Sodium 5mEq/kg/Day; Test type: Superiority; p = 0.57, Regression, Cox; Hazard Ratio (HR) = 0.62

ADVERSE EVENTS:
Time Frame: Through hospitalization stay, an expected average of 3 months.
Arm/Group | Sodium < 1mEq/kg/Day | Sodium 5mEq/kg/Day
All-Cause Mortality (participants affected / at risk) | 5/23 | 2/19
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/23 | 0/19

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT04035564/Prot_SAP_000.pdf